CLINICAL TRIAL: NCT00293813
Title: A Multicenter, Randomized Placebo Controlled Pilot MicroCT Study to Estimate the Effect of Treatment With Denosumab (AMG 162) and Alendronate Sodium in Postmenopausal Women With Low Bone Mineral Density
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20050179
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Post Menopausal; Osteoporosis; MicroCT; Amgen; denosumab; Extreme CT; XCT; Fosamax; Alendronate
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Alendronate; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 3 (Placebo Comparator): Placebo for denosumab and placebo for alendronate
  Interventions: Drug: Placebo
- 1 (Experimental): denosumab and placebo for alendronate
  Interventions: Drug: Denosumab
- 2 (Active Comparator): Placebo for denosumab and alendronate
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — Alendronate 70 mg PO QW
  Arms: 2
Drug: Denosumab — denosumab 60 mg SC q 6 mos
  Arms: 1
Drug: Placebo — Placebo for alendronate and placebo for denosumab
  Arms: 3

SUMMARY:
This study is structured to estimate the effect of denosumab, compared to placebo and alendronate, on several bone parameters.

ELIGIBILITY:
Key Inclusion Criteria:

* Postmenopausal, ambulatory women between 50 and 70 years old who are generally in good health.
* Must have low bone mineral density and meet specific eligibility criteria.

Key Exclusion Criteria:

-Subjects must not currently be receiving any medication that affects bone metabolism or have an underlying condition that affects their ability to take alendronate or receive denosumab.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Seeman E, Delmas PD, Hanley DA, Sellmeyer D, Cheung AM, Shane E, Kearns A, Thomas T, Boyd SK, Boutroy S, Bogado C, Majumdar S, Fan M, Libanati C, Zanchetta J. Microarchitectural deterioration of cortical and trabecular bone: differing effects of denosumab and alendronate. J Bone Miner Res. 2010 Aug;25(8):1886-94. doi: 10.1002/jbmr.81. PMID 20222106
- [Background] Zebaze RM, Libanati C, Austin M, Ghasem-Zadeh A, Hanley DA, Zanchetta JR, Thomas T, Boutroy S, Bogado CE, Bilezikian JP, Seeman E. Differing effects of denosumab and alendronate on cortical and trabecular bone. Bone. 2014 Feb;59:173-9. doi: 10.1016/j.bone.2013.11.016. Epub 2013 Nov 22. PMID 24275677
- [Derived] Hu YJ, Chines A, Shi Y, Seeman E, Guo XE. The effect of denosumab and alendronate on trabecular plate and rod microstructure at the distal tibia and radius: A post-hoc HR-pQCT study. Bone. 2022 Jan;154:116187. doi: 10.1016/j.bone.2021.116187. Epub 2021 Sep 14. PMID 34530172
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Alendronate 70 mg QW: Alendronate 70 mg QW
- Denosumab 60 mg Q6M: Denosumab 60 mg Q6M
- Placebo: Placebo
Period: Overall Study
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M | Placebo
Started | 82 | 83 | 82
Completed | 69 | 74 | 74
Not Completed | 13 | 9 | 8
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Withdrawal by Subject | 7 | 4 | 4
Not completed — Lost to Follow-up | 3 | 2 | 3
Not completed — Noncompliance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M | Placebo | Total
Number analyzed (Participants) | 82 | 83 | 82 | 247
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (5.2) | 60.3 (5.9) | 60.8 (5.2) | 60.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 83 | 82 | 247
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cortical Thickness of Radius by XtremeCT Percent Change From Baseline at Month 12
Description: Cortical Thickness measured by XtremeCT.
Time Frame: 12 months
Population: Randomized subjects who receive at least 1 dose of investigational product and have a baseline and at least 1 post baseline evaluation before or at month 12. Last Observation Carried Forward used as imputation method. Summarised for actual treatment taken.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 73 | 75 | 79
Percent Change from Baseline | 2.4 [1.2 to 3.5] | 3.4 [2.2 to 4.5] | -.8 [-1.8 to .3]
Statistical Analysis 1: Comparison: Denosumab 60 mg Q6M vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 4.1, 95% CI [2.6 to 5.7]
Statistical Analysis 2: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 1, 95% CI [-.6 to 2.6]

2. Secondary Outcome: Cortical Thickness of Tibia by XtremeCT Percent Change From Baseline at Month 12
Description: Cortical Thickness measured by XtremeCT.
Time Frame: 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 73 | 78 | 79
Percent Change from Baseline | 4.9 [4 to 5.8] | 5.8 [5 to 6.7] | 1.4 [.6 to 2.3]

ADVERSE EVENTS:
Arm/Group | Placebo | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 5/83 | 5/81 | 2/83
Other Adverse Events (participants affected / at risk) | 78/83 | 77/81 | 76/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | Alendronate 70 mg QW (N=81) | Denosumab 60 mg Q6M (N=83)
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | Alendronate 70 mg QW (N=81) | Denosumab 60 mg Q6M (N=83)
Abdominal pain (Gastrointestinal disorders) | 3 | 9 | 2
Abdominal pain upper (Gastrointestinal disorders) | 8 | 10 | 5
Constipation (Gastrointestinal disorders) | 12 | 13 | 15
Diarrhoea (Gastrointestinal disorders) | 9 | 10 | 3
Dyspepsia (Gastrointestinal disorders) | 7 | 9 | 5
Nausea (Gastrointestinal disorders) | 6 | 5 | 6
Vomiting (Gastrointestinal disorders) | 5 | 6 | 3
Bronchitis (Infections and infestations) | 11 | 11 | 9
Influenza (Infections and infestations) | 15 | 10 | 14
Nasopharyngitis (Infections and infestations) | 14 | 8 | 10
Pharyngitis (Infections and infestations) | 1 | 7 | 6
Urinary tract infection (Infections and infestations) | 5 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 10 | 10
Dizziness (Nervous system disorders) | 4 | 4 | 6
Headache (Nervous system disorders) | 9 | 12 | 6
Paraesthesia (Nervous system disorders) | 2 | 4 | 5
Breast mass (Reproductive system and breast disorders) | 3 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 6
Hypertension (Vascular disorders) | 6 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.